CLINICAL TRIAL: NCT01126021
Title: Using Technology to Promote Mental Acuity
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Carnegie Mellon University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS09-634
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-12

CONDITIONS: Mental Acuity
Keywords: Senior citizens; mental acuity; memory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Active Comparator): Given access to mental exercises but receives no rewards for use.
  Interventions: Behavioral: No incentives
- Atomistic (Experimental): Each individual is awarded for his or her individual participation
  Interventions: Behavioral: Financial incentives
- Altruistic (Experimental): Participants are paired and rewarded according to the other individual's participation.
  Interventions: Behavioral: Financial incentives
- Team-based (Experimental): Teams compete against each other and receive rewards according to relative participation.
  Interventions: Behavioral: Financial incentives

INTERVENTIONS:
Behavioral: Financial incentives — Participants are eligible for incentives if they participate in at least 30 games per day.
  Arms: Altruistic; Atomistic; Team-based
Behavioral: No incentives — Participants will be given training and access to the software to participate in mental exercises but will not be given financial incentives for participation.
  Arms: Control

SUMMARY:
The study plans to test the effectiveness of behavioral economics based incentives to promote the daily use of computer programs designed to improve memory and mental acuity. Subjects will be recruited from the Pittsburgh metropolitan area. The primary objective is to determine the impact of structured financial incentives on the number of computer-based cognitive exercises completed during a 3 month intervention period.

ELIGIBILITY:
Inclusion Criteria:

* 55-80 years old

Exclusion Criteria:

* Unable to read or understand the informed consent form

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2010-05; Primary Completion 2011-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Number of activities completed | 6 weeks
  The number of memory and cognition enhancement activities played per day using the study provided software will be measured.
Performance on activities completed | 6 weeks
  Performance is measured by a scoring algorithm designed to estimate levels of memory, attention, cognitive control and processing speed.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Carnegie Mellon University, Pittsburgh, Pennsylvania

REFERENCES:
- See also: LDI Center for Health Incentives — http://www.med.upenn.edu/ldichi/